CLINICAL TRIAL: NCT04116684
Title: Digital Home Blood Pressure Monitoring in Type B Aortic Dissection Patients
Acronym: Dissect-BP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with patient enrollment and carrying out the study logistics due to COVID-19
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-723
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Aortic Dissection; Hypertension
Keywords: Withings Blood Pressure Monitor; Heart Rate; Ambulatory Blood Pressure
MeSH Terms: conditions — Aortic Dissection; Hypertension

STUDY DESIGN:
Intervention Model Description: 50 patients will be randomly assigned to standard of care home blood pressure monitoring while the other 50 patients will be randomized to Withings home digital blood pressure monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (digital BP monitoring) (Experimental): This group will receive a Withings digital BP monitor to transmit recordings to the study team who will make medication adjustments.
  Interventions: Device: Withings Digital Blood Pressure Monitor
- Standard of care BP monitoring (No Intervention): This group will use a standard BP cuff and record and transmit data to their medical team as instructed by their providers or if they are concerned.

INTERVENTIONS:
Device: Withings Digital Blood Pressure Monitor — This is a home digital blood pressure monitor that can transmit recordings via a user's smartphone.
  Arms: Intervention Group (digital BP monitoring)

SUMMARY:
The primary objective of this study is to determine the effectiveness of home digital blood pressure monitoring in aiding providers to maintain blood pressure within a therapeutic range in type B aortic dissection patients upon discharge from the hospital.

DETAILED DESCRIPTION:
Patients admitted to the Cleveland Clinic Main Campus with a diagnosis of type B aortic dissection or intramural hematoma who do not receive a surgical intervention during their index hospitalization, or planned intervention on follow up, and are discharged on medical therapy consisting of strict heart rate control and BP control will be included in the study. They will be either randomized to standard therapy to measure BP at home (standard of care) or intervention arm consisting of Withings Wireless Blood Pressure Monitor, which will transmit BP recordings from smartphone to MyChart/EPIC (test arm). All patients will first receive a 24 hour ambulatory monitor regardless of treatment assignment to establish baseline BP pattern. Following this patients randomized to intervention arm will utilize their Withings Blood Pressure Monitor. Providers on the study team will then adjust the patient's hypertensive medications to ensure their BP is below a systolic goal of 120 mmHg utilizing downloaded recordings available in the electronic medical record.

The primary clinical endpoint is the change in mean 24 hour systolic blood pressure between the start of the study and the end of the study period (4-week period). Secondary outcomes will include the number of patients able to achieve a therapeutic systolic blood pressure of 120 mmHg with both mean BP cuff and in office visit at end of 4 week period, increase in size as measured by computed tomography (CT) scan of the aorta, hospitalization or emergency room (ER) visits for symptoms from dissection or uncontrolled hypertension, hospitalization or ER visits for hypotension, all-cause mortality, and need for surgical intervention (open or endovascular).

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from Cleveland Clinic Main Campus with principal diagnosis of type B aortic dissection (defined as distal from left subclavian artery) who do not receive a surgical intervention during their hospitalization
* Arm Circumference of 9-17 inches

Exclusion Criteria:

* Patients who do not have a smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venugopal Menon, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Started | 3 | 1
Completed | 1 | 1
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Digital BP Monitoring) | Standard of Care BP Monitoring | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure at End of 4 Weeks
Description: Systolic Blood Pressure at end of 4 weeks as measured by 24 hour ambulatory cuff.
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis was performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mortality
Description: Individual incidence of death
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Surgical Intervention
Description: Surgical intervention (open or endovascular)
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospitalization or Emergency Room Visit for Uncontrolled Hypertension or Symptoms From Dissection
Description: Individual occurrence of hospitalization or Emergency Room visit for uncontrolled hypertension or symptoms from dissection
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hospitalization or Emergency Room Visit for Hypotension
Description: Individual occurrence of hospitalization or Emergency Room visit for Hypotension
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Increase in Size or Progression of Dissection as Measured on Cardiac CT
Description: Incidence of Increase in size or progression of dissection compared to baseline as measured on cardiac CT
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Questionnaire Describing Patient Experience in the Study
Description: Collection of answers to questionnaire describing patient experience in the study
Time Frame: 4 weeks
Population: Study terminated prematurely due to COVID-19 pandemic; no analysis has been performed.
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks and 4 weeks
Arm/Group | Standard of Care BP Monitoring | Intervention Group (Digital BP Monitoring)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04116684/Prot_SAP_000.pdf